CLINICAL TRIAL: NCT02796690
Title: Staphylococcus Aureus Nasal Carriage Among Technical Staff of a Teaching Hospital: An Unexpected Group at Risk of Colonization
Brief Title: Staphylococcus Aureus Nasal Carriage
Acronym: SANAC
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL16_0337
Record Dates: First submitted 2016-06-07; First posted 2016-06-13 (Estimated); Last update posted 2016-06-13 (Estimated); Status verified 2016-06

CONDITIONS: Nasal Carriage of Staphylococcus Aureus
Keywords: nasal carriage; Staphylococcus aureus; good hygiene practices
MeSH Terms: conditions — Staphylococcal Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group Methicillin susceptible Staphylococcus aureus (MSSA)
  Interventions: Other: nasal swabs will be collected
- Group methicillin resistant Staphylococcus aureus (MRSA)
  Interventions: Other: nasal swabs will be collected

INTERVENTIONS:
Other: nasal swabs will be collected — After formal consent, nasal swabs are collected for each participant. SA nasal carriage and its susceptibility to methicillin is determined using a rapid PCR technique (GenExpert, Cepheid). Each participant is asked to complete a short questionnaire regarding some demographic variables, smoking habits, long-term medication, sector of activity, and direct manipulation of the pathogen.

SUMMARY:
The repeated exposition to S. aureus is considered as a determining factor of acquisition of the nasal colonization. The healthcare professionals are regularly in touch with this pathogenic bacterium. Prevalence of the nasal carriage of S. aureus in this population was the object of several studies but little took into account the respect for the rules of good hygienic practice. The results of our previous study carried out during the international congress of staphylococci (ISSSI, Lyon in August 26-30th, 2012) showed an association between the work in a hospital environment and the increase of the risk of nasal carriage. On the contrary, the use of the hydro-alcoholic solutions had a protective effect against this carriage. However, sized of the health care population of our study was limited.

The goal of this study is to confirm our previous results on a larger cohort of healthcare professionals. The main objective is to estimate the prevalence of nasal carriage according to the professional category and by taking into account the degree of conformity with good hygiene practices including the use of hydro-alcoholic solutions.

ELIGIBILITY:
Inclusion Criteria:

- Employees with Consent.

Exclusion Criteria:

- Presence of contraindicating medical conditions preventing nasal swabing

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Employees of a teaching hospital in Lyon-France
Sampling Method: Non-Probability Sample
Enrollment: 310 (Actual)
Dates: Start 2014-04; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Rate of nasal carriage of Staphylococcus aureus (SA) among employees of a teaching hospital in Lyon-France according to professional exposure and compliance with good hygiene practices. | after 2 days

SECONDARY OUTCOMES:
Prevalence of nasal carriage of Staphylococcus aureus (SA) methicillin susceptible (MSSA) or methicillin resistant (MRSA) among employees of a teaching hospital in Lyon-France. | after 2 days
Presence or not of nasal carriage of Staphylococcus aureus (SA) among employees of a teaching hospital in Lyon-France at particular conditions as long medication intake and overweight. | after 2 days

CONTACTS AND LOCATIONS:
Overall Officials: François Vandenesch, Pr, Principal Investigator — National Reference Center for Staphylococci
Locations (1):
- National Reference Center for Staphylococci, 59 boulevard Pinel, Bron, France